CLINICAL TRIAL: NCT01304459
Title: Vancomycin Serum Concentrations in Pediatric Oncology Patients Under Intensive Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, GLAUCIA TORIBIO FINOTI SEIXAS, MD, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Other Study IDs: UTI/IOP 01/11; 1913/10 (Other: CEP UNIFESP)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational protocol to analyse routine vancomycin serum levels of patients under intensive care and to obtain percentage of patients that achieve therapeutic values.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized pediatric oncology patients
* Patients under vancomycin treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric oncology patients on intensive care unit for treatment of infections.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Apoio ao Adolescente e à Criança com Câncer, São Paulo, São Paulo, Brazil